CLINICAL TRIAL: NCT05346380
Title: Near-Infrared Perfusion During Minimally Invasive Thoracic Surgery
Brief Title: Near-Infrared Perfusion During Minimally Invasive Thoracic Surgery Download
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Olympus (Industry)
Responsible Party: Principal Investigator, Christopher R. Morse, M.D., Principal Investigator MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020P000835
Record Dates: First submitted 2022-02-11; First posted 2022-04-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Lung Neoplasms; Esophageal Lesion
MeSH Terms: conditions — Lung Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: The treatment arms are separated by type of surgery. Arm 1 is esophagectomy, Arm 2 is segmentectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- During Minimally Invasive Pulmonary Segmentectomy (Group 2) (Experimental)
  Interventions: Device: Olympus VE2 NIR Imaging System; Drug: Indocyanine green
- During Minimally Invasive Esophagectomy (Group 1) (Experimental)
  Interventions: Device: Olympus VE2 NIR Imaging System; Drug: Indocyanine green

INTERVENTIONS:
Device: Olympus VE2 NIR Imaging System — A prospective, (NSR), single-center feasibility study of the Olympus VE2 NIR Imaging System to assess perfusion using NIR during minimally invasive esophagectomy or pulmonary segmentectomy based on treatment arm.
Drug: Indocyanine green — intravenous delivery of low-dose 0.15 mg/kg of ICG combined with Olympus VE2 NIR Imaging System to assess perfusion using NIR during minimally invasive esophagectomy or pulmonary segmentectomy based on treatment arm

SUMMARY:
This will be a prospective, (NSR), single-center feasibility study of the Olympus VE2 NIR Imaging System to assess perfusion using NIR during minimally invasive esophagectomy and pulmonary segmentectomy. The aims of the study are:

1. To utilize NIR intraoperative imaging with the Olympus VE2 NIR Imaging System to: i. Characterize gastric conduit perfusion during esophagectomy and, ii. Identify segmental anatomy during sublobar pulmonary resection (segmentectomy) after intraoperative, intravenous delivery of low-dose 0.15 mg/kg of ICG.

DETAILED DESCRIPTION:
Current Surgical Approaches to Thoracic Malignancies are Imperfect: Thoracic malignancies are among the most deadly cancers diagnosed across the world. Non-small cell lung cancer (NSCLC) remains the number one cause of cancer related mortality in the United States and across the world. Esophageal cancer is the second most common thoracic malignancy, and is the fastest growing malignancy in the United States. Together, these 2 tumor types account for more an annual mortality of 150,000 in the United States alone. For patients with stage I and stage II disease, surgery provides the best opportunity for long-term survivorship for both malignancies; however, operative intervention is associated with significant morbidity and upwards of 20% of patients have complications.

As with surgery involving other body cavities, safe oncologic resection of thoracic tumors involves a careful understanding of the arterial blood flow to tissues that are to be (1) resected and (2) left behind. Despite the importance of these considerations, there remains very few tools to help the surgeon with this assessment. Two examples of these clinical dilemmas involve (1) pulmonary artery delineation during pulmonary segmentectomy and (2) conduit assessment during esophagectomy. Consequences of improper perfusion assessment can involve a variety of complications such as leak, stricture, abscess, or unnecessary resection.

This protocol describes a tool to address these unmet needs. More specificall, this non-significant risk study will assess feasibility of the Olympus VISERA ELITE II Near-infrared (VE2 NIR) Imaging System (Olympus Medical Systems Corp., Tokyo, Japan to intraoperatively assess perfusion during (1) pulmonary segmentectomy and (2) gastric conduit perfusion during esophagectomy by detecting systemically delivered indocyanine green (ICG). The VE2 NIR Imaging system has obtained 510k clearance from the US FDA for blood flow and related tissue perfusion.

Indocyanine Green (ICG): Indocyanine green is a water-soluble, NIR fluorophore with a molecular weight of 774.9 kDA. When intravenously delivered, ICG binds to plasma albumin thus creating a circulating nanoparticle. The main mechanism of excretion is hepatic as the liver excretes more than 80% of the available ICG in less than 24 hours. ICG is the most intensively studied NIR contrast agent and was approved by the United States Food and Drug Administration (FDA) for human administration in 1958. As a fluorophore, ICG has a peak absorption wavelength of 805 nm and a peak emission wavelength of 830 nm. ICG is inexpensive, non-toxic and readily available, making it an ideal contrast agent for intraoperative NIR imaging. The FDA specifically approves ICG for cardiac output, hepatic function and ophthalmic angiography.

Previous clinical data pertaining to ICG-based NIR imaging of gastric conduit perfusion at the time of esophagectomy: Esophagectomy remains a mainstay of multi-modality therapy for esophageal cancer. During esophagectomy, the diseased esophagus is resected and the remaining portion of the stomach (gastric conduit) is brought through the chest where it is anastomosed to either the thoracic or cervical esophagus. Anastomotic and conduit complications significantly contribute to morbidity and mortality associated with esophagectomy. Adequate vascular perfusion of the gastric conduit is vital to avoid these complications. To date, conduit viability is assessed intraoperatively by surgeon observational assessment, which is subjective. Thoracic surgeons are in desperate need of new technologies that can better assess tissue perfusion and ischemia of the gastric conduit. One such technique is the use of intraoperative NIR imaging with ICG to directly assess these parameters.

To date, hundreds of patients have been involved studies of NIR imaging with ICG to assess gastric conduit perfusion. In this approach, low dose ICG (2.5mg-25mg) is intravenously delivered and imaging of the neo-esophageal conduit commences 30 seconds later. In a review of over 420 patients undergoing this approach, this NIR signal was found to be reproducible, with no observed toxicity. Authors reported benefits of NIR imaging in identifying otherwise non-detectable transverse vessels between the terminal arcade and the short gastric arteries. Perhaps more convincing, in a propensity score matched study involving over 214 subjects, patients undergoing esophagectomy with the addition of NIR with ICG were found to have a 3-fold decrease (p=0.03) in anastomotic complications when compared to those undergoing traditional esophagectomy. Our goal is to utilize the Olympus VE2 NIR Imaging System with ICG to evaluate gastric conduit perfusion during minimally invasive esophagectomy.

Previous clinical experiences involving ICG-based NIR imaging to assess segmental anatomy during pulmonary resection: According to 2019 National Comprehensive Cancer Network (NCCN) Guidelines, the gold-standard treatment of resectable malignant pulmonary lesions requires anatomic resection (pneumonectomy, lobectomy or segmentectomy) with lymph node sampling. For patients with lesions larger than 2cm, lobectomy or pneumonectomy is typical. However, for lesions less than 2cm segmentectomy has been demonstrated to provide equivalent oncologic outcomes while also preserving functional lung parenchyma. Despite parenchymal sparing benefits, anatomic delineation of pulmonary segments is challenging and inaccurate. Current segmentectomy approaches involve careful clamping of those segmental airways supplying lung parenchyma involved with tumor burden, followed by insufflation of the ipsilateral lung. Using this approach, the non-clamped (cancer free) lung inflates while the clamped (lung to be resected) remains atelectatic. The surgeon then resects the "non-inflated" lung. Because of collateral ventilatory networks among alveoli and obstructive changes associated with lung cancer, lines of demarcation between these lung areas is often unclear. Inaccurate resection along segmental planes may result in retention of devascularized tissue, inadequate surgical margins, or incomplete clearing of draining lymphatic pathways.

Given challenges associated with current segmentectomy approaches, many groups have begun utilizing intraoperative NIR imaging with ICG to better demarcate segmental anatomy. To date, thousands of patients across dozens of institutions have utilized this method. In this approach, low dose ICG (ranging from 10-50mg) is delivered intravenously after clamping segmental pulmonary artery. Within minutes of ICG delivery, unclamped (healthy) parenchyma demonstrates a strong NIR signal which is detected using a modified thoracoscope, while the clamped (to be resected) tissue remains dark. In these studies reporting toxicity, there were minimal side effects from the ICG delivery. Our goal is to utilze the Olympus VE2 NIR Imaging System when used with ICG to assess segmental perfusion anatomy during minimally invasive sublobar pulmonary segmentectomy.

ELIGIBILITY:
Inclusion Criteria:

-Subject has a suspicious lung lesion for which a minimally invasive segmentectomy is planned -OR- sub-ject has an esophageal lesion for which an esophagectomy is planned -

* Subject is 18 years of age or older
* Subject is willing and able to provide informed consent

Exclusion Criteria:

* Subject is not eligible for surgical resection as determined by the treating physician
* Subject has known or suspected allergy to Iodine, shellfish or intravenous contrast

  * Subject is not eligible or considered high risk for surgical resection as determined by pre-operative spirometry
  * Subject is female and of childbearing age who is currently pregnant or who is planning to become pregnant within the study
  * Subject is unable and unwilling to provide informed consent
  * Subject has liver disease or is taking drugs impact liver metabolism.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
To utilize NIR intraoperative imaging with the Olympus VE2 NIR Imaging System for esophagectomy patients. | During surgery
  Fluorescent intensity, visualization of the intersegmental plane with NIR imaging, image quality will all be ranked by the surgeon as "below standard, average, or good" compared to the standard of care as they identify segmental anatomy during sublobar pulmonary resection (segmentectomy) after intraoperative, intravenous delivery of low-dose 0.15 mg/kg of ICG.
To utilize NIR intraoperative imaging with the Olympus VE2 NIR Imaging System for segmentectomy patients. | During surgery
  Fluorescent intensity, visualization of the intersegmental plane with NIR imaging, image quality will all be ranked by the surgeon as "below standard, average, or good" compared to the standard of care as they identify esophageal anatomy during esophagectomy after intraoperative, intravenous delivery of low-dose 0.15 mg/kg of ICG.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Morse, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Sharing device and surgical data with Olympus, however no PHI will be shared.

REFERENCES:
- [Background] DeLong JC, Kelly KJ, Jacobsen GR, Sandler BJ, Horgan S, Bouvet M. The benefits and limitations of robotic assisted transhiatal esophagectomy for esophageal cancer. J Vis Surg. 2016 Sep 8;2:156. doi: 10.21037/jovs.2016.09.01. eCollection 2016. PMID 29078542
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402